CLINICAL TRIAL: NCT01951066
Title: Diabetic Macular Edema Treated With Ozurdex (DMEO)
Acronym: DMEO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Peter A Campochiaro, MD, Professor of Ophthalmology and Neuroscience, Johns Hopkins University
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DMEO-001
Record Dates: First submitted 2013-09-20; First posted 2013-09-26 (Estimated); Results first posted 2016-08-01 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-08

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (dexamethasone implant/anti-VEGF) (Experimental): Patients in group 1 received an injection of an dexamethasone implant at baseline followed by PRN anti-VEGF injections after crossover at week 16.
  Interventions: Drug: Dexamethasone Implant; Drug: Anti-VEGF injection
- Group 2 (anti-VEGF/dexamethasone implant) (Experimental): Patients in group 2 received prn anti-VEGF injections followed by injection of a dexamethasone implant after crossover at week 16.
  Interventions: Drug: Dexamethasone Implant; Drug: Anti-VEGF injection

INTERVENTIONS:
Drug: Dexamethasone Implant — Patients will receive a single injection of a dexmethasone implant
Drug: Anti-VEGF injection — Patients will receive PRN injections of an anti-VEGF agent

SUMMARY:
To measure various pro-permeability factors in the aqueous humor of patients with persistent/recurrent diabetic macular edema

DETAILED DESCRIPTION:
Patients with Diabetic Macular Edema (DME) are increasingly being treated with molecules targeting vascular endothelial factor (VEGF). One potential advantage of a dexamethasone implant over specific VEGF antagonists is that steroids suppress production of multiple pro-permeability factors.

Our primary objective is to measure the pro-permeability factors in the aqueous humor of patients with persistent/recurrent macular edema despite prior treatment with anti-VEGF agents at baseline and at 1, 2, 3, and 4 months after intraocular injection of a dexamethasone implant.

ELIGIBILITY:
Inclusion Criteria:

* • Signed informed consent and authorization of use and disclosure of protected health information

  * Age more than or equal to 18 years
  * Diagnosis of diabetic macular edema
  * Intraretinal or subretinal fluid in the macula determined by Spectralis OCT
  * Best corrected visual acuity score in the study eye of 20/30 to 20/400 inclusive (Snellen equivalents using the ETDRS protocol at a distance of 4 meters)
  * In the opinion of the investigator, decreased vision in the study eye is due to foveal thickening from DME and not from other obvious causes of decreased vision
  * Persistent or recurrent edema despite prolonged treatment with an anti-VEFG agent

Exclusion Criteria:

* • Scatter laser photocoagulation or macular photocoagulation within 3 months of study entry in the study eye

  * Intraocular surgery in the study eye within 3 months of study entry
  * Use of intraocular or periocular injection of steroids in the study eye (e.g., triamcinolone) within 4 months of study entry
  * Previous use of an anti-VEGF drug within 1 month of study entry
  * Yttrium-Aluminum-Garnet (YAG) laser capsulotomy within 1 month of study entry
  * Any condition that the investigator believes would pose a significant hazard to the subject if investigational therapy were initiated.
  * Inability to comply with study or follow up procedures
  * History of glaucoma. (Patients who have undergone filtration surgery may be included)
  * Patients with active or suspected ocular or periocular infection, including most viral diseases of the cornea and conjunctiva, including active epithelial herpes simplex keratitis (dendritic keratitis), vaccinia, varicella, mycobacterial infections, and fungal diseases.
  * Aphakic eyes with rupture of the posterior lens capsule.
  * Eyes with ACIOL and rupture of the posterior lens capsule.
  * Patients with hypersensitivity to dexamethasone or to any other components of the product

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Campochiaro, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Wilmer Eye Institute, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (Baseline to Week 16)
Arm/Group | Group 1 (Dexamethasone Implant/Anti-VEGF) | Group 2 (Anti-VEGF/Dexamethasone Implant)
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Intervention (Week 16 to Week 32)
Arm/Group | Group 1 (Dexamethasone Implant/Anti-VEGF) | Group 2 (Anti-VEGF/Dexamethasone Implant)
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 61.8 [47 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Baseline Intraretinal Fluid [Number; unit: participants]
  Mild | 3
  Moderate | 14
  Severe | 3
Mean Disease Duration [Mean (Full Range); unit: Months] | 48.1 [3 to 132]
Prior Anti-VEGF injections [Mean (Full Range); unit: Injections] | 13.3 [0 to 56]
Prior Intraocular Steroids [Number; unit: participants] | 5
Prior Laser [Number; unit: participants]
  Grid Laser | 6
  Scatter Laser Photocoagulation | 6
Baseline Best Corrected Visual Acuity [Mean (Full Range); unit: ETDRS Score] — The Best Corrected Visual Acuity (BCVA) was measured using the Early Treatment of Diabetic Retinopathy Study (ETDRS) Score. Patient can have an ETDRS score ranging from 5 to 100. A higher ETDRS Score represents better visual acuity.
  ETDRS Score | 56.1 [30 to 74]
Baseline Central Subfield Thickness [Mean (Full Range); unit: Microns] — The Central Subfield Thickness (CST) was measured using Spectralis OCT machine.
  Microns | 464.3 [280 to 779]

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Change in Level of Propermeability Factors With Change in Edema After Treatment With a Dexamethasone Implant or Anti-VEGF Agent
Description: Changes in propermeability factor levels were correlated with changes in edema using the person correlation coefficient (this was calculated using data from all time points).
Time Frame: 1, 2, 3, and 4 months after injection of a dexamethasone implant or anti-VEGF agent
Measure: Number; unit: Pearson correlation coefficient (r)
Groups:
- Dexamethasone Implant: Patients received an injection of an dexamethasone implant
- Anti-VEGF Agent: Patients received PRN injections of an Anti-VEGF agent
Arm/Group | Dexamethasone Implant | Anti-VEGF Agent
Number analyzed (Participants) | 20 | 20
Pearson correlation coefficient (r)
  IGF-BP1 | 0.47 | 0.059
  Prolactin | 0.45 | 0.369
  MMP-9 | 0.45 | 0.29
  EG-VEGF | 0.43 | -0.004
  Endostatin | 0.41 | 0.189
  Angiopoietin-2 | 0.40 | 0.229
  IGF-BP3 | 0.36 | 0.435
  Persephin | 0.35 | 0.114
  MIP-1a | 0.34 | -0.107
  THSP-2 | 0.33 | 0.064
  HGF | 0.31 | 0.226
  IL-8 | 0.30 | -0.184
  CXCL16 | 0.29 | 0.027

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 4/20
Other Adverse Events (participants affected / at risk) | 11/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=20)
Cataract progression (Eye disorders) | 1
Emergency room visit because of a possible seizure (Nervous system disorders) | 1
Mitral valve repair surgery (Cardiac disorders) | 1
Endophthalmitis (Eye disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=20)
Steroid injection in the hip due to arthritis (Musculoskeletal and connective tissue disorders) | 1
Racing of heart (Cardiac disorders) | 1
Foot Infection (Musculoskeletal and connective tissue disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Vision loss (Eye disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Patient had a fall (General disorders) | 2
Increased Intraocular pressure (Eye disorders) | 1
Eye soreness (Eye disorders) | 1
Bruising of eyelid (Eye disorders) | 1
Blood transfusion due to severe anemia (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other